CLINICAL TRIAL: NCT05088954
Title: Effect of Metabolic Syndrome on Outcomes of Transforaminal Epidural Steroid Injection Treatment in Patients With Chronic Lumbar Radiculopathy
Brief Title: Effect of Metabolic Syndrome on Outcomes of Transforaminal Epidural Steroid Injection Treatment in Chronic Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2021.1040
Record Dates: First submitted 2021-10-21; First posted 2021-10-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Herniated Disk Lumbar; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: transforaminal epidural steroid injection
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients diagnosed with metabolic syndrome (Active Comparator)
  Interventions: Procedure: transforaminal epidural steroid injection
- Patients without a diagnosis with metabolic syndrome (Active Comparator)
  Interventions: Procedure: transforaminal epidural steroid injection

INTERVENTIONS:
Procedure: transforaminal epidural steroid injection — In the transforaminal approach, a small amount of drug is injected into the epidural space, and in previous studies, reduction in pain and improvement in functionality were found in patients with lumbar radicular pain in the short and medium term.

SUMMARY:
Transforaminal epidural steroid injection (TFESI) has been increasingly preferred in patients who can not benefit from conservative approach in the treatment of lumbosacral radiculopathic pain due to lumbar disc herniation. The aim of our study is to evaluate the effect of metabolic syndrome on the treatment results of transforaminal epidural steroid injection in patients with chronic radicular low back pain due to lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* lumbar radiculopathy due to lumbar disc herniation, unresponsive to conservative treatments, duration of pain is at least 3 months, Patients aged 18 and above

Exclusion Criteria:

* the cases when fluoroscopy or epidural injection is contraindicated (coagulation disorders, pregnancy etc...), to have a history of lumbar spinal surgery, inflammatory diseases (rheumatoid arthritis, spondyloarthropathy), spinal infection or malignancy, systemic infection, Spondylolisthesis or spinal stenoz at the involved or adjacent segments, allergies to local anesthetics, contrast dyes or steroids, Refusal of a patient, History of prior lumbar spine surgery, presence of hip pathology (avascular necrosis, congenital hip dislocation etc...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of Successful Response | 6 months
  The primary outcome measure of our study is successful response (>50% reduction in NRS)

SECONDARY OUTCOMES:
Numerical Rating Scale | 6 months
  The patient is asked to give a score between 1 and 10 to explain the pain level. The change in NRS compared to the baseline was measured at the outpatient visit.
Istanbul Low Back Pain Disability Index (ILBPDI) | 6 months
  Istanbul Low Back Pain Disability Index (ILBPDI) is a scale developed to evaluate functional disability in patients with chronic low back pain, scoring 18 subjects. The change in ILBPDI compared to the baseline was measured at the outpatient visit.
Short Form 12 (SF-12) | 6 months
  Short Form 12 (SF-12) is a quality of life assessment scale consisting of 8 sub-dimensions and 12 items. The change in SF-12 compared to baseline is measured at the outpatient visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)